CLINICAL TRIAL: NCT01652729
Title: A Randomized, Long-Term, Open-Label, 3-Arm, Multicenter Study to Compare the Glycemic Effects, Safety, and Tolerability of Exenatide Once Weekly Suspension to Sitagliptin and Placebo in Subjects With Type 2 Diabetes Mellitus
Brief Title: Comparison Study of the Glycemic Effects, Safety, and Tolerability of Exenatide Once Weekly Suspension to Sitagliptin and Placebo in Subjects With Type 2 Diabetes Mellitus
Acronym: DURATION-NEO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCB120; MB001-004 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Type 2
Keywords: Diabetes, Type 2, exenatide, Sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exenatide once weekly suspension (Experimental): Exenatide once weekly suspension 2mg subcutaneous injection
  Interventions: Drug: Exenatide once weekly suspension
- Sitagliptin 100mg (Active Comparator): Overencapsulated Sitagliptin 100mg oral tablet once daily
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo oral capsule once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide once weekly suspension
  Arms: Exenatide once weekly suspension
Drug: Sitagliptin
  Arms: Sitagliptin 100mg
Drug: Placebo — Placebo oral capsule once daily
  Arms: Placebo

SUMMARY:
To compare the effect on glycemic control (HbA1c) of exenatide suspension administered once weekly to that achieved by sitagliptin or placebo administered once daily for 28 weeks in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed with type 2 diabetes mellitus
* HbA1c of 7.1% to 11.0%, inclusive, at screening
* Has stable body weight, i.e., not varying by >3% for at least 3 months prior to screening
* Fasting plasma glucose concentration <280 mg/dL (15.5 mmol/L) at screening
* Body mass index of <45 kg/m2 at screening
* Has been treated with a stable regimen of ≥1500 mg/day metformin for a minimum of 2 months prior to Visit 1 (Screening)

Exclusion Criteria:

* History of pancreatitis or triglycerides >=500 mg/dL
* Medullary carcinoma or multiple endocrine neoplasia (MEN2) or a family history of either
* History of renal transplantation, or is currently receiving renal dialysis, or has an estimated creatinine clearance <50 mL/min
* Active cardiovascular disease
* Presence or history of severe congestive heart failure
* Central nervous system disease, including epilepsy
* Liver disease
* History of severe gastrointestinal diseases
* Clinically significant malignant disease
* Repeated severe hypoglycemia within the last 6 months
* Any exposure to exenatide (BYETTA® or BYDUREON™) or any GLP-1 analog
* Any DPP-4 inhibitor within 3 months prior screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ohman, Study Chair — AstraZeneca
Locations (53):
- United States (53):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Buena Park, California
  - Research Site, Chino, California
  - Research Site, Chula Vista, California
  - Research Site, Encinitas, California
  - Research Site, Greenbrae, California
  - Research Site, Los Angeles, California
  - Research Site, North Hollywood, California
  - Research Site, Walnut Creek, California
  - Research Site, West Hills, California
  - Research Site, Boca Raton, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Orange, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Oxon Hill, Maryland
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Hartsdale, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Clayton, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Franklin, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Yukon, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Greer, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Reseach Site, Rapid City, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Carrolton, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burke, Virginia
  - Research Site, Spokane, Washington

REFERENCES:
- [Derived] Guja C, Frias JP, Suchower L, Hardy E, Marr G, Sjostrom CD, Jabbour SA. Safety and Efficacy of Exenatide Once Weekly in Participants with Type 2 Diabetes and Stage 2/3 Chronic Kidney Disease. Diabetes Ther. 2020 Jul;11(7):1467-1480. doi: 10.1007/s13300-020-00815-z. Epub 2020 Apr 18. PMID 32306296
- [Derived] Gadde KM, Vetter ML, Iqbal N, Hardy E, Ohman P; DURATION-NEO-2 study investigators. Efficacy and safety of autoinjected exenatide once-weekly suspension versus sitagliptin or placebo with metformin in patients with type 2 diabetes: The DURATION-NEO-2 randomized clinical study. Diabetes Obes Metab. 2017 Jul;19(7):979-988. doi: 10.1111/dom.12908. Epub 2017 Mar 17. PMID 28205322
- See also: BCB120_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2733&filename=BCB120_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomly assigned across 3 treatment groups (exenatide, sitagliptin, and placebo) in a ratio of 3:2:1, with randomization stratified by screening HbA1c stratum (< 9% or 9%).
Groups:
- Experimental: Exenatide: Exenatide once weekly suspension 2mg subcutaneous injection
- Active Comparator: Sitagliptin: Sitagliptin 100mg oral tablet once daily
- Placebo Comparator: Placebo: Placebo oral tablet once daily
Period: Overall Study
Arm/Group | Experimental: Exenatide | Active Comparator: Sitagliptin | Placebo Comparator: Placebo
Started | 182 (One subject was enrolled twice at different sites. He was randomized to exenatide at both sites.) | 122 | 61
Modified Intent-to-Treat | 181 (All randomized subjects who received at least one dose of study drug.) | 122 | 61
Treated | 181 (All subjects who received at least one dose of study medication even if not randomized.) | 122 | 61
Evaluable | 143 (Subjects who completed study procedures to Week 24 or beyond and had adequate study drug exposure) | 91 | 43
Meal Test Subjects | 60 | 41 | 20
Meal Test Evaluable | 44 (ITT subjects who ate >=75% of meal and did not miss 2-hour postprandial glucose measures at V3 and 8) | 31 | 15
Completed | 155 (The double-enrolled subject's reasons for withdrawal were LTFU and PV. Only PV is shown below.) | 109 | 47
Not Completed | 27 | 13 | 14
Not completed — Withdrawal by Subject | 14 | 7 | 7
Not completed — Adverse Event | 4 | 0 | 3
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 6 | 6 | 3
Not completed — Administrative | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Exenatide | Active Comparator: Sitagliptin | Placebo Comparator: Placebo | Total
Number analyzed (Participants) | 181 | 122 | 61 | 364
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (9.82) | 54.3 (9.01) | 53.4 (9.48) | 53.7 (9.49)
Age, Customized [Number; unit: Participants]
  <65 years | 154 | 106 | 54 | 314
  >=65 years | 27 | 16 | 7 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 56 | 24 | 172
  Male | 89 | 66 | 37 | 192
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 148 | 98 | 50 | 296
  Black or African American | 24 | 18 | 7 | 49
  Asian | 9 | 2 | 3 | 14
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Other | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 111 | 77 | 32 | 220
  Not Hispanic or Latino | 70 | 45 | 29 | 144
Weight [Mean (Standard Deviation); unit: kg] | 89.15 (21.413) | 88.09 (20.282) | 88.95 (20.136) | 88.76 (20.778)
Baseline HbA1c [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.42 (0.997) | 8.50 (1.043) | 8.50 (1.043) | 8.46 (1.018)
HbA1c Stratum [Number; unit: participants]
  < 9.0% | 125 | 83 | 42 | 250
  >= 9.0% | 56 | 39 | 19 | 114
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 178.0 (46.64) | 176.9 (42.50) | 172.8 (44.31) | 176.8 (44.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Hemoglobin) From Baseline to Week 28
Description: Absolute change in HbA1c from baseline (Day 1, Visit 3) to Week 28/Study Termination (Visit 11). Hypothesis testing on the primary endpoint followed a serial gated procedure with all tests carried out at a 2-sided significance level of 0.05 to protect the family-wise error rate. These tests were conducted sequentially, and are presented in the statistical analysis section below in the order in which they were performed; each test was the gatekeeper of later tests.
Time Frame: Baseline to Week 28
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Experimental: Exenatide | Active Comparator: Sitagliptin | Placebo Comparator: Placebo
Number analyzed (Participants) | 181 | 122 | 61
percentage of total hemoglobin | -1.13 (0.1093) | -0.75 (0.1324) | -0.40 (0.1945)
Statistical Analysis 1: Comparison: Experimental: Exenatide vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 0.0010, mixed model for repeated measure; MMRM includes treatment, baseline HbA1c (<9% or ≥9%), week of visit and treatment by visit interaction as fixed factors, and subject random effect; LS Mean Difference = -0.72, 95% CI 2-sided [-1.15 to -0.30], Standard Error of Mean 0.2167
Statistical Analysis 2: Comparison: Experimental: Exenatide vs Active Comparator: Sitagliptin; Test type: Superiority or Other; p = 0.0209, mixed model for repeated measure; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.38, 95% CI 2-sided [-0.70 to -0.06], Standard Error of Mean 0.1638
Statistical Analysis 3: Comparison: Active Comparator: Sitagliptin vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 0.1347, mixed model for repeated measure; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.34, 95% CI 2-sided [-0.79 to 0.11], Standard Error of Mean 0.2278

2. Secondary Outcome: Percentage of Subjects Achieving HbA1c <7% at Week 28
Description: Percentage of subjects achieving HbA1c target values of < 7.0% at Week 28/Study Termination.
Time Frame: Baseline to Week 28
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug.
Measure: Number; unit: percentage of subjects
Arm/Group | Experimental: Exenatide | Active Comparator: Sitagliptin | Placebo Comparator: Placebo
Number analyzed (Participants) | 181 | 122 | 61
percentage of subjects
  Baseline Yes | 3.3 | 1.6 | 3.3
  Baseline No | 96.7 | 98.4 | 96.7
  Week 28 Yes | 43.1 | 32.0 | 24.6
  Week 28 No | 56.9 | 68.0 | 75.4
Statistical Analysis 1: Comparison: Experimental: Exenatide vs Active Comparator: Sitagliptin; Percentage of Subjects Achieving HbA1c <7% at Week 28; Test type: Superiority or Other; p = 0.0489, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Experimental: Exenatide vs Placebo Comparator: Placebo; Percentage of Subjects Achieving HbA1c <7% at Week 28; Test type: Superiority or Other; p = 0.0103, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change in Fasting Plasma Glucose Concentrations From Baseline to Week 28
Description: The change in fasting plasma glucose concentrations from baseline (Day 1) to Week 28/Study Termination.
Time Frame: Baseline to Week 28
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Experimental: Exenatide | Active Comparator: Sitagliptin | Placebo Comparator: Placebo
Number analyzed (Participants) | 181 | 122 | 61
mg/dL | -21.3 (3.864) | -11.3 (4.617) | 9.6 (7.097)
Statistical Analysis 1: Comparison: Experimental: Exenatide vs Active Comparator: Sitagliptin; Test type: Superiority or Other; p = 0.0924, mixed model for repeated measure; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -10.1, 95% CI 2-sided [-21.8 to 1.7], Standard Error of Mean 5.960
Statistical Analysis 2: Comparison: Experimental: Exenatide vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 0.0001, mixed model for repeated measure; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -30.9, 95% CI 2-sided [-46.7 to -15.1], Standard Error of Mean 8.037

4. Secondary Outcome: Change in Body Weight (kg) From Baseline to Week 28
Description: The change in body weight (kg) from baseline (Day 1) to Week 28/Study Termination.
Time Frame: Baseline to Week 28
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Experimental: Exenatide | Active Comparator: Sitagliptin | Placebo Comparator: Placebo
Number analyzed (Participants) | 181 | 122 | 61
kg | -1.12 (0.2592) | -1.19 (0.3134) | 0.15 (0.4767)
Statistical Analysis 1: Comparison: Experimental: Exenatide vs Active Comparator: Sitagliptin; Test type: Superiority or Other; p = 0.8625, mixed model for repeated measure — Nominal p-value; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.07, 95% CI 2-sided [-0.73 to 0.87], Standard Error of Mean 0.4058
Statistical Analysis 2: Comparison: Experimental: Exenatide vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 0.0198, mixed model for repeated measure — Nominal p-value; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.27, 95% CI 2-sided [-2.34 to -0.20], Standard Error of Mean 0.5419

5. Secondary Outcome: Change in 2-hour Postprandial Glucose Concentrations From Baseline to Week 16 (Visit 8)
Description: The change in 2-hour postprandial plasma glucose from baseline (Day 1) to Visit 8 (Week 16) was analyzed using a general linear model including treatment, and baseline HbA1c stratum (< 9% or ≥ 9%) as fixed factors, and the baseline 2-hour postprandial plasma glucose concentrations as a covariate.
Time Frame: Baseline to Week 16
Population: Meal Test Evaluable Population: The Meal Test Evaluable Population consists of all modified ITT subjects who participated in the meal test, consumed at least 75% of the standardized meal and had no missing 2-hour postprandial glucose measurements at both Visit 3 (Day 1) and Visit 8 (Week 16), and have adequate study drug exposure.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Experimental: Exenatide | Active Comparator: Sitagliptin | Placebo Comparator: Placebo
Number analyzed (Participants) | 44 | 31 | 15
mg/dL | -59.57 (10.48) | -23.61 (13.04) | -38.68 (16.98)
Statistical Analysis 1: Comparison: Experimental: Exenatide vs Active Comparator: Sitagliptin; Test type: Superiority or Other; p = 0.0248, general linear model — Nominal p-value; Includes treatment and baseline HbA1c (< 9% or ≥ 9%) as fixed factors, and baseline 2-hour postprandial plasma glucose concentrations as a covariate; LS Mean Difference = -35.96, 95% CI 2-sided [-67.23 to -4.68], Standard Error of Mean 15.71
Statistical Analysis 2: Comparison: Experimental: Exenatide vs Placebo Comparator: Placebo; Test type: Superiority or Other; p = 0.2914, general linear model — Nominal p-value; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = -20.89, 95% CI 2-sided [-60.02 to 18.25], Standard Error of Mean 19.66

ADVERSE EVENTS:
Arm/Group | Experimental: Exenatide | Active Comparator: Sitagliptin | Placebo Comparator: Placebo
Serious Adverse Events (participants affected / at risk) | 5/181 | 0/122 | 2/61
Other Adverse Events (participants affected / at risk) | 31/181 | 2/122 | 4/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Exenatide (N=181) | Active Comparator: Sitagliptin (N=122) | Placebo Comparator: Placebo (N=61)
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain Stem Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Exenatide (N=181) | Active Comparator: Sitagliptin (N=122) | Placebo Comparator: Placebo (N=61)
Nausea (Gastrointestinal disorders) | 16 (18) | 2 (2) | 0 (0)
Injection Site Nodule (General disorders) | 14 (19) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less